CLINICAL TRIAL: NCT05014776
Title: A Phase 2 Study of the Safety, Efficacy, and Immune Response of CRS-207, Pembrolizumab, Ipilimumab, and Tadalafil in Patients With Previously Treated Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of CRS-207, Pembrolizumab, Ipilimumab, and Tadalafil in Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Lustgarten Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2180; IRB00291762 (Other: Johns Hopkins Medical Institution); 5P01CA247886 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pembrolizumab; Ipilimumab; CRS-207; Tadalafil; Immunotherapy; Anti-PD-1; Anti-CTLA-4; Adenocarcinoma; Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Carcinoma | interventions — Tadalafil; pembrolizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207 (Experimental)
  Interventions: Drug: Tadalafil; Drug: Pembrolizumab; Drug: Ipilimumab; Drug: CRS-207

INTERVENTIONS:
Drug: Tadalafil — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Tadalafil (20 mg) will be administered orally every day on days 3-21 for cycles 1-6.
  Other Names: CIALIS®
Drug: Pembrolizumab — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on Day 1 of cycles 1-6.
  Other Names: KEYTRUDA®
Drug: Ipilimumab — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Ipilimumab (50mg) will be administered IV on Day 1 of Cycles 1, 3, and 5.
  Other Names: YERVOY®
Drug: CRS-207 — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 [1 × 10^9 colony forming units (CFU) in 100ml NS] will be administered IV on Day 2 of Cycles 1-6.

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of tadalafil, pembrolizumab, ipilimumab, and CRS-207 in subjects with metastatic pancreatic adenocarcinoma who have progressed after at least 1 prior chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Have histologically or cytologically proven adenocarcinoma of the pancreas.
* Have previously treated metastatic disease.
* Have radiographic disease progression.
* Patients with the presence of at least one measurable tumor lesion.
* Patient's acceptance to have a tumor biopsy at baseline and on
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Known history or evidence of brain metastases.
* Had chemotherapy, radiation, or biological cancer therapy within the last 14 days.
* Have received an investigational agent or device within the last 28 days.
* Had surgery within the last 28 days.
* Expected to require any other form of systemic or localized cancer therapy while on study.
* Have received a vaccine within the last 14 days (7 days for the COVID vaccine) or received a live vaccine within the last 30 days.
* Have received steroids within the last 14 days.
* Use more than 4 g/day of acetaminophen.
* Use of organic nitrates.
* Use of guanylate cyclase (GC) stimulators such as riociguat.
* Consumption of substantial amounts of alcohol (≥5 units/day)
* Use of strong or moderate cytochrome P450 3A4 (CYP3A4) inhibitor or inducer.
* Patients on immunosuppressive agents within the last 7 days
* Known allergy to both penicillin and sulfa.
* Severe hypersensitivity reaction to any monoclonal antibody.
* History of severe hypersensitivity to tadalafil.
* Have implant(s) or device(s) that has not and cannot be easily removed.
* Have artificial joints or implanted medical devices that cannot be easily removed.
* Have any evidence of clinical or radiographic ascites.
* Have significant and/or malignant pleural effusion
* Uncontrolled intercurrent illness.
* Subjects with active, known or suspected autoimmune disease.
* Have a tissue or organ allograft, including corneal allograft.
* Have been diagnosed HIV, Hepatitis B or C positive.
* Is on supplemental home oxygen.
* Has an unhealed surgical wound or ulcer, or a bone fracture considered non-healing.
* Has clinically significant heart disease
* Prior history of non-arterial ischemic optic retinopathy.
* History of significant hypotensive episode requiring hospitalization within 6 months.
* Has insufficient peripheral vein access.
* Is unwilling or unable to follow the study schedule for any reason.
* Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2026-04-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bever, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207
Started (Started = enrolled and received at least one dose of study drug) | 17
Completed (Completed = Received 1 course (6 cycles) of treatment) | 3
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using Response Evaluation Criteria for Solid Tumors (RECIST 1.1)
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. Participants who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders. Participants who discontinue for other reasons prior to their first dose of study drug will not included in the analysis.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Number of Participants Experiencing Drug-Related Adverse Events (AEs) Requiring Treatment Discontinuation
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 12 months. All-cause mortality was evaluated for up to 16 months.
Arm/Group | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207
All-Cause Mortality (participants affected / at risk) | 16/17
Serious Adverse Events (participants affected / at risk) | 12/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207 (N=17)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Biliary Obstruction (Gastrointestinal disorders) | 2 (2)
Bowel Obstruction (Gastrointestinal disorders) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 1 (2)
Disease Progression (General disorders) | 11 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Tadalafil, Pembrolizumab, Ipilimumab, CRS-207 (N=17)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (10)
Ascites (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bloating (Gastrointestinal disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (2)
Chills (General disorders) | 17 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Creatinine increased (Investigations) | 3 (4)
Dark stool (Gastrointestinal disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dizziness (Nervous system disorders) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema (General disorders) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 7 (8)
Fever (General disorders) | 15 (37)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Floaters (Eye disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (9)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (13)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypotension (Vascular disorders) | 5 (7)
Hypothyroidism (Endocrine disorders) | 2 (2)
COVID Infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 10 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (6)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (7)
Skin and subcutaneous tissue disorders - Lump (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Weight gain (Investigations) | 3 (3)
Weight loss (Investigations) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05014776/Prot_SAP_000.pdf